CLINICAL TRIAL: NCT05125068
Title: A Phase 2a, Multicenter, Open-Label Study to Evaluate the Safety and Efficacy of AT-1501 in Patients With IgA Nephropathy
Brief Title: Safety and Efficacy of AT-1501 in Patients With IgA Nephropathy (IgAN)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: An administrative decision was made to terminate the AT-1501-N205 study. This voluntary business-related decision was not related to the safety of tegoprubart (AT-1501). Available safety data demonstrated tegoprubart to be safe and well tolerated.
Sponsor: Eledon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-1501-N205; 2021-004795-34 (EudraCT Number); U1111-1269-7356 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: IgA Nephropathy; IgAN
Keywords: IgA Nephropathy; IgAN; AT-1501; CD40L; Monoclonal antibody; Proteinuria; eGFR; UPCR
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): AT-1501 10mg/kg Arm A will receive 10 mg/kg of AT-1501 every 3 weeks for up to 93 weeks for a total of 32 infusions.
  Interventions: Drug: AT-1501
- Arm B (Experimental): AT-1501 5mg/kg Arm B will receive 5 mg/kg of AT-1501 every 3 weeks for up to 93 weeks for a total of 32 infusions
  Interventions: Drug: AT-1501

INTERVENTIONS:
Drug: AT-1501 — AT-1501 monoclonal antibody targeting CD40L given as an IV infusion

SUMMARY:
This is a phase 2a, multicenter, open-label study designed to evaluate the safety and efficacy of AT-1501 in patients with biopsy proven IgAN and at least 0.75 g/24 hours of protein in their urine at the time of screening.

DETAILED DESCRIPTION:
Phase 2a, multicenter, open-label study designed to evaluate the safety and efficacy of AT-1501 in patients with biopsy proven IgAN and at least 0.75 g/24 hours of protein in their urine at the time of Screening. Up to 42 eligible patients will receive one of 2 doses of AT-1501. All patients are scheduled to receive AT-1501 by intravenous infusion every 3 weeks for approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Biopsy proven IgAN
3. Urine protein ≥ 0.75g/24 hours at Screening despite optimization with ACE inhibitors or angiotensin receptor blockers (ARB)
4. eGFR ≥ 45 mL/min per 1.73 m2 or eGFR < 45 mL/min per 1.73 m2 and ≥ 30 mL/min per 1.73 m2 with a kidney biopsy within 2 years of Screening showing < 50% tubulointerstitial fibrosis
5. Agree to comply with contraception requirements during and for 90 days after study completion.

Exclusion Criteria:

1. Any secondary IgAN as defined by the investigator
2. Patients who have undergone a kidney transplant
3. Any history of kidney disease other than IgAN
4. Any history of diabetes (Type 1 or Type 2)
5. Seated blood pressure > 140 mmHg (systolic) or > 90 mmHg (diastolic) at the Screening Visit. Patients must be on a stable dose and regimen of an ACE inhibitor or ARB for at least 90 days
6. Pregnancy or breastfeeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Efficacy - change in participants UPCR | Up to 24 weeks
  The change in 24-hour urine protein to creatinine ratio (UPCR) from baseline to 24 weeks
Safety- Number of participants with treatment related adverse events | Through study completion, an average of 100 weeks
  Incidence of serious adverse events (SAEs), treatment-emergent adverse events (TEAEs), and AEs of special interest (AEoSI)

SECONDARY OUTCOMES:
Change in eGFR slope | Baseline- 96 weeks
  The change in eGFR slope from baseline to 96 weeks
Change in urine protein excretion (mg/mg) | Up to 96 weeks
  The change in urine protein excretion over time
Development of Anti drug Antibodies (ADAs) | Up to 96 weeks
  The percentage of participants who develop ADAs

OTHER OUTCOMES:
Exploratory- Change in baseline serum biomarkers | Through study completion, an average of 100 weeks
  The change in serum biomarkers from baseline to completion of study

CONTACTS AND LOCATIONS:
Locations (26):
- Australia (3):
  - Liverpool Hospital, Liverpool, South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Western Health, St Albans, Victoria
- Croatia (2):
  - University Hospital Centre Sisters of Charity, Zagreb
  - University Hospital Dubrava Zagreb, Zagreb
- Malaysia (5):
  - University Malaya Medical Centre (UMMC), Kuala Lumpur, Kuala Lumpur WP
  - Hospital Tengku Ampuan Afzan (HTAA), Kuantan, Pahang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Kajang, Kajang, Selangor
  - Hospital Serdang, Kajang, Selangor
- New Zealand (2):
  - Waikato Hospital, Hamilton
  - Hawke's Bay Hospital, Hastings
- University of Santo Tomas Hospital, Sampaloc, Manila, Philippines
- Poland (2):
  - Medical University of Bialystok UI, Bialystok
  - Specjalistyczne Centrum Medyczne, SCM Spółka, Krakow
- Spain (4):
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen de la Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Sri Lanka (2):
  - National Hospital of Sri Lanka, Colombo
  - Sri Jayawardanepura General Hospital, Nugegoda
- Thailand (4):
  - Prince of Songkla University, Dusit, Bangkok
  - Chulalongkorn University, Pathum Wan, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
- Kings College Hospital, Camberwell, United Kingdom